CLINICAL TRIAL: NCT06622018
Title: Effect of Seashell Nanoparticles and Gluma Desensitizer on Sensitivity of Teeth Prepared for Intra Coronal Restorations as Well as Micromorphology of The Treated Dentin Surfaces
Brief Title: Effect of Seashell Nanoparticles and Gluma Desensitizer on Sensitivity of Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hoda Fathy El gendy, Specialist of Dental Medicine, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hoda El Gendy
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-01

CONDITIONS: Teeth Sensitivity; Treated Dentin Surfaces
MeSH Terms: conditions — Dentin Sensitivity | interventions — gluma desensitizer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Control Group) (Placebo Comparator): About 11 patients with hypersensitive teeth of no treatment materials used
  Interventions: Procedure: Seashell Nanoparticles and Gluma Desensitizer
- Group B(Seashell Nanoparticles Group) (Active Comparator): About 11 patients with hypersensitive teeth faced treatment by sea shell nanoparticles
  Interventions: Procedure: Seashell Nanoparticles and Gluma Desensitizer
- Group C (Gluma Group) (Active Comparator): About 11 patients with hypersensitive teeth faced treatment by Gluma
  Interventions: Procedure: Seashell Nanoparticles and Gluma Desensitizer

INTERVENTIONS:
Procedure: Seashell Nanoparticles and Gluma Desensitizer — Evaluation the effect of Seashell Nano Particles and Gluma desensitizer on sensitivity of the teeth for Intra coronal restoration at different times
  Other Names: Micromorphology

SUMMARY:
Tooth hypersensitivity is characterized by a transient short and sharp pain originating from exposed dentin in response to thermal, dehydrating, tactile, osmotic, and chemical stimuli. Tooth sensitivity after cementation of complete coverage crowns, is a rather common event since much of the protecting enamel is removed during preparation and a large area of dentin is exposed.

Dentin contains up to two million tubules per cm2, which corresponds approximately to the surface area of most crown preparations. It is well known that such dentin wounds respond to mechanical, osmotic, or thermal stimulation with pain. This phenomenon is commonly example by the hydrodynamic theory of Brannstrom.

DETAILED DESCRIPTION:
The extent and duration of post cementation hypersensitivity has been related to number of factors, mainly associated with preparation trauma. However, research reports confirm potential effects of luting agents used and leakage of bacteria and bacterial products from the oral cavity along the margins of restorations, especially as a response to poorly fitting temporary restorations. Apparently, a relationship exists between the time interval during which the temporary restoration is in place and post cementation sensitivity.

Gluma Desensitizer is a combination of glutaraldehyde and HEMA (Hydroxy Ethyl Methacrylate). Glutaraldehyde causes amino acids and proteins to coagulate in dentinal tubules and is an effective disinfectant. HEMA can be effective in sealing of dentinal tubules.

Gluma does not interfere with dentin bonding systems but its glutaraldehyde component can damage the gingiva after long term exposure. HEMA can cause contact dermatitis and it can actually perforate latex gloves and must be used with caution, hence, the use of rubber dam is advised in such cases .

HEMA is soluble in water allowing it to penetrate deep into dentinal tubules however, the effect is reversible and HEMA gradually loses its effect allowing the dentinal tubules to again became exposed.

Hydroxyapatite powder is one such material that exhibits excellent bioactive properties and striking similarities to dental hard tissues can be achieved from two different sources. Synthetic and natural (biologic) hydroxyapatite.HAP can be produced from Coral Seashells, eggshells and also from body fluids.

Recently, the use of waste materials to synthesize HAP has received great response from many researchers across the world. This idea gives an innovation to produce a new valuable product from the waste materials such as seashell.Seashell consists of high source of calcium that can act as calcium precursor. Some researcher found that the content of calcium carbonate (CaCO3) in seashell is approximately between 98 and 99 %.

The word seashell is often used to mean only the shell of a marine mollusk. Using seashell as source of calcium carbonate (CaCO3) to produce calcite nanoparticle is meaningful for both environmental protection and biomedical application. Seashell is with the natural ceramic structure are similar to human bone and tooth structure.

The conversation of macroparticles into nanoparticles resulted in larger surface area increasing the reactivity of nanoparticles and hence, it's efficacy. Nanoparticles have widespread use due to their superior properties and are being investigated extensively in recent years due to their advantages.Nano -sized materials can enter dentinal tubules of 2 -3 µm in diameter, easily occluding the dentinal tubules

ELIGIBILITY:
Inclusion Criteria:

* For patient Age between 25 and 40 years and no gender reference.
* For the teeth Absence of pulpal exposure, RCT treatments, fracture and free of extensive caries (The amount of caries that can be removed during the preparation is acceptable

Exclusion Criteria:

* -For patients Use of desensitizing substances or drug like antihistamines, antidepressant 6 weeks before or during the study.

Requiring antibiotic prophylaxes or cortico-steriod therapy.

-For teeth Tooth hypersensitivity prior to tooth preparation (like, abrasion or attration).

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Desnsetizing agent Hypersensitivity | from 0 hours to two weeks
  Evaluation of the treated patients from hypersensitivity of the application of desnsetizing agent ( gluma and nanasaesheall) by using VAS score (from 0 to 10) as 0 is mean no sensitivity while 10 is the worst.

SECONDARY OUTCOMES:
Dentinal tubule occlusion | from 0 hours to two weeks
  Ability of the materials to induce dentinal tubule occlusion using SEM

CONTACTS AND LOCATIONS:
Overall Officials: Osama Saleh Abd El Ghani, Professor, Study Chair — Al-Azhar Faculty of Dental Medicine for girls
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided